CLINICAL TRIAL: NCT01648257
Title: A Single-center, Randomized, Open-label, Crossover Study to Assess the Relative Bioavailability of New Formulations of GSK1265744 in Healthy Adult Subjects
Brief Title: Relative Bioavailability Study of GSK1265744 Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116585
Record Dates: First submitted 2012-07-19; First posted 2012-07-24 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Infections, Human Immunodeficiency Virus and Hepatitis
Keywords: healthy subjects; relative bioavailability; HIV; GSK1265744
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK1265744 Na Salt Tablets (Experimental): Subjects will receive single dose of GSK1265744 sodium salt (30 mg) tablet on Day 1 of the respective period per randomized sequence, orally in fasted condition, with 240 milliliter (mL) of water.
  Interventions: Drug: GSK1265744 Na Salt Tablets
- GSK1265744 Free Acid Nanomilled Capsules (Experimental): Subjects will receive single dose of GSK1265744 free acid nanomilled (30 mg) capsule on Day 1 of the respective period per randomized sequence, orally in fasted condition, with 240 mL of water.
  Interventions: Drug: GSK1265744 Free Acid Nanomilled Capsules
- GSK1265744 Free Acid Micronized Capsules (Experimental): Subjects will receive single dose of GSK1265744 free acid micronized (30 mg) capsule on Day 1 of the respective period per randomized sequence, orally in fasted condition, with 240 mL of water.
  Interventions: Drug: GSK1265744 Free Acid Micronized Capsules

INTERVENTIONS:
Drug: GSK1265744 Na Salt Tablets — Each tablet contains 30 mg of GSK1265744 sodium salt and excipients.
  Arms: GSK1265744 Na Salt Tablets
Drug: GSK1265744 Free Acid Nanomilled Capsules — Each capsule contains 30 mg of nanomilled and spray dried GSK1265744 free acid, blended with excipients.
  Arms: GSK1265744 Free Acid Nanomilled Capsules
Drug: GSK1265744 Free Acid Micronized Capsules — Each capsule contains 30 mg of micronized GSK1265744 free acid, blended with excipients.
  Arms: GSK1265744 Free Acid Micronized Capsules

SUMMARY:
This is a single-center, randomized, open-label, balanced, 3 way crossover study (3 periods) in healthy adult subjects. During each period, subjects will receive a single dose of GSK1265744 oral formulation in the fasted state and serial PK sampling for up to 168 hours (8 days) and safety assessments will be performed. Each period will be separated by a washout period of at least 14 days and a follow-up visit will occur 10 to 14 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin =< 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinically significant abnormality or laboratory parameter outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 64 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, bilateral salpingo-oophorectomy or hysterectomy; postmenopausal defined in the protocol; or child-bearing potential and agrees to use one of the contraception methods listed in the protocol.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* Body weight >= 50 kilogram (kg) for men and >= 45 kg for women and body mass index (BMI) within the range 18.5 to 31.0 kg/ (meters squared) m^2 (inclusive).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* History of regular alcohol consumption within 6 months of the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new investigational chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive urine human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* The subject's systolic blood pressure is outside the range of 90-140 millimeters of mercury (mmHg), or diastolic blood pressure is outside the range of 45 to 90 mmHg.
* History of clinically significant cardiovascular disease.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Composite of PK parameters following single oral dose administration of GSK1265744 | For 168 hours post dose (36 days)
  Plasma GSK1265744 PK parameters: area under the concentration-time curve (AUC) from time zero (pre-dose) extrapolated to infinite time AUC(0-infinity); AUC from time zero to time t, AUC(0-t), and maximum observed concentration, Cmax.

SECONDARY OUTCOMES:
Composite of PK parameters following single oral dose administration of GSK1265744 | For 168 hours post each dose of GSK1265744 (36 days)
  Following plasma GSK1265744 PK parameters will be evaluated: concentration at 24 hour post-dose (C24), terminal phase half-life (t1/2), lag time before observation of drug concentrations in sampled matrix (tlag), time of occurrence of Cmax (tmax), percentage of AUC(0-infinity) obtained by extrapolation (%AUCex), apparent clearance following oral dosing (CL/F).
Safety and tolerability as assessed by the collection of adverse events | 50 days
Safety and tolerability as assessed by change from baseline in clinical laboratory tests | 50 days
  Clinical laboratory tests include hematology, clinical chemistry, urinalysis tests.
Safety and tolerability as assessed by change from baseline in electrocardiogram (ECG) | 50 days
Safety and tolerability as assessed by change from baseline in vital signs | 50 days
  Vital sign measurements will include systolic and diastolic blood pressure and pulse rate.
Safety and tolerability as assessed by the collection of concurrent medication. | 50 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States